CLINICAL TRIAL: NCT01674491
Title: Effects of Black Soy Peptide Supplementation on Blood Pressure and Oxidative Stress:A Randomized Controlled Trial
Brief Title: Effects of Black Soy Peptide Supplementation on Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BPS_201106
Record Dates: First submitted 2012-08-10; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4.5g/day black soy peptide (Experimental): 4.5 g/day, 8weeks
  Interventions: Dietary Supplement: black soy peptide
- placebo (Placebo Comparator): similar appearance to the black soy peptide tablet, 8 weeks
  Interventions: Dietary Supplement: black soy peptide

INTERVENTIONS:
Dietary Supplement: black soy peptide — black soy peptide: 4.5g/day for 8 weeks

SUMMARY:
Black soy peptides have been shown to possess properties that may decrease blood pressure. To examine the effects of black soy peptides supplementation on blood pressure and oxidative stress in subjects with pre-hypertension or stage I hypertension.

DETAILED DESCRIPTION:
Trial participants included men and women aged 30 to 65 years who had an average systolic blood pressure (SBP) between 130 to 159 mmHg, average diastolic blood pressure (DBP) between 80 to 99 mmHg, or both, based on an average of six measurements during two screening visits. Participants were supplied with 84 pouches of placebo (casein) or black soy peptide (3 pouches/day) at 0-week and at 4-week visits. Test group subjects received pouches containing black soy peptides (4.5 g/day total soy peptides for 8 weeks). The control group received pouches containing casein that had a similar appearance to the black soy peptide tablet. During the intervention, we instructed study participants to continue their current food intake patterns and lifestyles so that total energy intake and energy expenditure would be constant during the course of trial. Participants brought back unconsumed pouches at their 4- and 8-week follow-up visits. The dietitian counted the number of returned pouches, and we used this to assess the participants' adherence to their assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* Average systolic blood pressure (SBP) between 130 to 159 mmHg
* Average diastolic blood pressure (DBP) between 80 to 99 mmHg, or both, based on an average of six measurements during two screening visits

Exclusion Criteria:

* Previous diagnosed clinical hypertension
* Self-reported use of anti-hypertensive medication
* Abnormal liver or renal function
* History of cardiovascular disease, cancer, thyroid or pituitary disease, or any other serious life-threatening illness that required regular medical treatment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change from baseline in Systolic blood pressure at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Diastolic blood pressure at 8 weeks | 8 weeks
change from baseline in plasma malondialdehyde at 8 weeks | 8 weeks
change from baseline in Urinary 8-epi-prostaglandin F2 at 8 weeks | 8 weeks
change from baseline in Renin at 8 weeks | 8 weeks
Change from baseline in angiotensin-converting enzyme at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D, Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomic, Seoul, South Korea